CLINICAL TRIAL: NCT05875948
Title: A Single-blind, Phase 2, Multi-center, Randomized Study to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of the R2R01 Plus Terlipressin Versus Terlipressin Alone in Patients With Hepatorenal Syndrome - Acute Kidney Injury
Brief Title: Study to Evaluate R2R01 Plus Terlipressin Versus Terlipressin Alone in Patients With Hepatorenal Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: River 2 Renal Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: R2R01-HRS-201
Record Dates: First submitted 2023-05-01; First posted 2023-05-25 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-05

CONDITIONS: Hepatorenal Syndrome; Acute Kidney Injury
Keywords: HRS-AKI; HRS; Renal Failure; Kidney Failure; Single-blind; Open-Label; Phase 2; R2R01
MeSH Terms: conditions — Hepatorenal Syndrome; Acute Kidney Injury; Renal Insufficiency | interventions — Terlipressin

STUDY DESIGN:
Intervention Model Description: A. An Open-Label Safety Run-In Part with 3 Cohorts of patients, followed by
  B. A Single-Blind Placebo-Controlled Randomized Part with two Cohorts of patients treated in parallel, and
  C. An Open-Label Terlipressin Non-Responder Cohort.
Who Masked: Participant
Masking Description: Patients in Cohorts 4 and 5 will be blinded to study treatment. Patients randomized to Cohort 4 will receive terlipressin and R2R01. Patients randomized to Cohort 5 will receive terlipressin and R2R01-matching placebo in the same schedule as Cohort 4. Study staff and Investigators will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- An Open-Label Safety Run-In Part (Experimental): Three initial cohorts (Cohort 1, N=3 patients, Cohorts 2 and 3, N=6 patients, each) will be treated with an open-label combination of terlipressin and R2R01 to ascertain the safety of the combination therapy.
  A Safety Review Committee (SRC) will review the safety of Cohort 1 patients based on the adverse events and laboratory abnormalities up until Day 14, prior to the start of recruitment of Cohort 2 patients, as well as the safety of Cohorts 1 and 2 patients up until Day 14 prior to the start of recruitment of Cohort 3 patients.
  Data from all Cohorts 1, 2, and 3 patients up until Day 14 will be reviewed by the SRC before starting the randomized part of the study (Cohorts 4 and 5), so that the SRC can decide and confirm the most appropriate R2R01 dose schedule for patients in Cohorts 4 and 5. Patients enrolled in Cohorts 1, 2, or 3 will remain in their Cohort until study completion (Day 90) or study discontinuation.
  Interventions: Drug: R2R01; Drug: Terlipressin
- Single-blind Placebo-controlled Randomized period (Placebo Comparator): After conclusion of the open-label safety run-in part, and after the SRC has determined the appropriate R2R01 dose schedule, approximately 80 patients will receive terlipressin and be randomized 1:1 to either R2R01 (Cohort 4) or placebo (Cohort 5).
  At randomization, patients will be stratified by the presence of systemic inflammatory response syndrome (SIRS), since patients with SIRS have shown a better response to terlipressin than patients without SIRS.
  Interventions: Drug: R2R01; Drug: Terlipressin
- An Open-Label Terlipressin Non-Responder Cohort (Experimental): In Cohort 5, if patients do not respond to terlipressin, they must discontinue Cohort 5. After discontinuation, they will be allowed to enter Cohort 6 (Terlipressin Non-Responder Part) to receive R2R01 with the same dosing and schedule as that for Cohort 4. No patient from any Cohort other than Cohort 5 will be allowed to enter Cohort 6.
  Interventions: Drug: R2R01; Drug: Terlipressin

INTERVENTIONS:
Drug: R2R01 — Pharmaceutical form: sterile 2R vials containing 10 mg of R2R01.
Drug: Terlipressin — In the US, terlipressin is supplied as a sterile, preservative-free, lyophilized, white-to- off-white powder for intravenous (IV) administration. Each vial contains 0.85 mg Terlivaz, equivalent to 1 mg terlipressin acetate, and 10.0 mg mannitol. Terlivaz requires reconstituting in saline (5mL).
  In the EU, terlipressin is supplied in a clear glass vial with 5 ml of injection solution, containing 1 mg terlipressin acetate corresponding to 0.85 mg terlipressin.

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of R2R01 combined with terlipressin as compared to terlipressin alone in the treatment of patients with HRS-AKI

DETAILED DESCRIPTION:
This is a phase 2 randomized, single-blind, placebo-controlled, two group, multicenter trial preceded by a safety run-in, in patients with Hepatorenal Syndrome (HRS) - Acute Kidney Injury (HRS-AKI).

The study consists of:

A. an Open-Label Safety Run-In Part with 3 Cohorts of patients, followed by

B. a Single-Blind Placebo-Controlled Randomized Part with two Cohorts of patients treated in parallel, and

C. an Open-Label Terlipressin Non-Responder Cohort.

All patients in all Cohorts will be treated with terlipressin, administered as a slow intravenous (IV) bolus 1 mg over 2 minutes every 6 hours (h) to be increased if clinically appropriate to 2.0 mg every 6 h. Terlipressin dosing should continue up to 24 h after achievement of an HRS response (either Partial or Full) based on Serum Creatinine (SCr)/AKI stage or up to day 14.

For those Cohorts where terlipressin will be administered combined with R2R01 (i.e., Cohorts 1, 2, 3, 4, and 6), the first R2R01 administration will commence immediately following the first terlipressin administration. Like terlipressin treatment, R2R01 dosing should continue up to 24 h after achievement of an HRS response (either Partial or Full) based on SCr/AKI stage or up to day 14.

All patients in all Cohorts will be followed for up to 90 days after the first dose of study drug.

This study will be conducted across approximately 25 centers in EU, UK, US, and Canada.

The screening period will occur within 14 days prior to the first dose administration.

The treatment duration is up to 14 days with a follow-up period of approximately 76 days.

The expected total duration of study participation is up to 15 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to communicate well with the Investigator, understands and is willing to comply with all requirements of the study, and understands and signs the written informed consent form (ICF).
2. At least 18 years of age.
3. Cirrhosis and ascites.
4. AKI stage 2 or 3. AKI defined by any of the following: 1) increase in SCr (SCr) ≥ 0.3 mg/dl (or ≥ 26.5 micromolar/L) within 48 h, or 2) increase ≥ 50% in baseline SCr, which is known or presumed to have occurred within the prior seven days.
5. QLY SCr ≥ to 1.5 mg/dl.
6. No sustained improvement in renal function (less than 20% decrease in SCr and SCr => 1.5 mg/dL) after 48 h of diuretic withdrawal and the beginning of plasma volume expansion with albumin.
7. Female patients as well as female partners of male patients must be willing to avoid pregnancy for the duration of the study (>90 days).

Exclusion Criteria:

1. Significant co-morbidities that in the opinion of the Investigator would preclude study participation.
2. QLY SCr level > 5 mg/dL.
3. AKI stage 1.
4. ACLF stage 3.
5. Model for End-Stage Liver Disease (MELD) score >35.
6. At least one event of large volume paracentesis (LVP) > 4 Liters in the last 4 days before enrollment.
7. Current or recent (within 4 weeks) treatment with nephrotoxic drugs (e.g., aminoglycosides, amphotericin, cyclosporine, NSAIDS (e.g., ibuprofen, naproxen, celecoxib), significant exposure to radiographic contrast agents (large doses or multiple injections of iodinated contrast media).
8. Shock (hypovolemic-, cardiogenic-, or vasodilatory/distributive shock) with mean arterial blood pressure (MAP) ≤70 mmHg or systolic blood pressure ≤90 mmHg along with hypoperfusion.
9. Sepsis or uncontrolled bacterial infection (e.g., persisting bacteremia, persisting ascitic fluid leucocytosis, fever, increasing leucocytosis with vasomotor instability) as measured with the quick sepsis-related organ dysfunction assessment (qSOFA) score.
10. Fewer than two days of anti-infective therapy for documented or suspected infection.
11. Superimposed acute liver injury induced by drugs, herbal preparation or dietary supplements, with the exception of alcoholic hepatitis.
12. Estimated life expectancy less than 5 days.
13. Hypoxia (<90%) or worsening respiratory symptoms.
14. Proteinuria > 500 mg/day.
15. Tubular epithelial casts, heme granular casts.
16. Haematuria or microhaematuria (more than 50 red blood cells per high power field).
17. Abnormal renal ultra-sonography unless there is a known chronic structural disease (e.g., diabetic or hypertensive nephropathy).
18. Current or recent (within 4 weeks) renal replacement therapy (RRT).
19. Severe cardiovascular and pulmonary diseases including, but not limited to, unstable angina, pulmonary edema, congestive heart failure requiring increasing doses of drug therapy, persisting symptomatic peripheral vascular disease, or any other cardiovascular disease judged by the Investigator to be severe.
20. Transjugular intra-hepatic systemic shunt (TIPS) unless it is known to be non-functioning or occluded.
21. Ongoing use of vasopressors, unless used for only 48 h before screening; in this case a wash-out period of 8 h before enrollment will be necessary. Patients receiving midodrine and octreotide may be enrolled but treatment must be discontinued prior to enrollment.
22. Known allergy or hypersensitivity to terlipressin or other component of the study treatment.
23. Subject is not suitable to participate in the study for any reason (including, but not limited to co-morbidities, history of non-compliance with study visits, procedures, or drug administration) in the opinion of the Investigator.
24. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study unless they agree to use highly effective contraception.
25. Males who have no sterilization history and whose female partners have child-bearing potential must agree to use a highly effective method of contraception during the period from the time of signing the informed consent form (ICF) through 90 days after the last dose of study drug. A male patient must agree to immediately inform the Investigator if his partner becomes pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation Criteria - Treatment Emergent Adverse Events (TEAEs) | From first dose of study drug to 30 days post last dose
  Safety and tolerability will be assessed by occurrence of TEAEs. Outcome will be reported as the count of participant experiencing TEAEs.
Safety Evaluation Criteria - Change in Weight | Change from screening through Day 30
  Safety and tolerability will be assessed by change in body weight
Safety Evaluation Criteria - Vital Signs - Respiration Rate | Change from screening through Day 30
  Safety and tolerability will be assessed by change in respiration rate
Safety Evaluation Criteria - Vital Signs - Body Temperature | Change from screening through Day 30
  Safety and tolerability will be assessed by change in body temperature
Safety Evaluation Criteria - Vital Signs - Continuous pulse oximetry (SpO2) | Change from baseline through Day 30
  Safety and tolerability will be assessed by change in SpO2
Safety Evaluation Criteria - Vital Signs - Systolic Blood Pressure (SBP) | Change from screening through Day 30
  Safety and tolerability will be assessed by change in SBP
Safety Evaluation Criteria - Vital Signs - Diastolic Blood pressure (DBP) | Change from screening through Day 30
  Safety and tolerability will be assessed by change in DBP
Safety Evaluation Criteria - Vital Signs - Heart Rate (HR) | Change from screening through Day 30
  Safety and tolerability will be assessed by change in Heart Rate (HR)
Safety Evaluation Criteria - ECGs - PR interval | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
Safety Evaluation Criteria - ECGs - RR interval | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
Safety Evaluation Criteria - ECGs - QRS duration | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
Safety Evaluation Criteria - ECGs - QT interval | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
Safety Evaluation Criteria - ECGs - QTcF interval | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
Safety Evaluation Criteria - ECGs - QTcB interval | Change from screening to Day 14 or hospital discharge
  Safety and tolerability will be assessed by occurrence of ECGs
The incidence of Responders | 90 days
  The incidence of Responders (Established HRS reversal defined as patients with a Full or Partial HRS response (based on SCr/AKI stage) AND are alive without Renal Replacement Therapy (RRT) for at least 30 days after the first dose of study medication), evaluated separately as two different outcome groups and combined. In case of recurrence and retreatment during the first 30 days, the second treatment period will be evaluated for response

SECONDARY OUTCOMES:
Mortality Rate | 30, 60, 90 days
  Number of patients who died at day 30, 60, and 90.
Liver Transplant Rates | 30, 60, 90 days
  Number of patients undergoing a liver transplant at day 30, 60, and 90.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Piedmont Healthcare, Inc, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No